CLINICAL TRIAL: NCT00058149
Title: A Phase III, Randomized Study of Gemcitabine (Fixed-Dose Rate Infusion) and Oxaliplatin (NSC 266046) Versus Gemcitabine (Fixed-Dose Rate Infusion) Versus Gemcitabine (30-Minute Infusion) in Pancreatic Carcinoma
Brief Title: Gemcitabine With or Without Oxaliplatin in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000287015; ECOG-6201
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2004-04

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine and oxaliplatin use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them in different ways may kill more tumor cells. It is not yet known whether gemcitabine is more effective with or without oxaliplatin in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of gemcitabine with or without oxaliplatin in treating patients who have locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival of patients with locally advanced or metastatic pancreatic cancer treated with prolonged infusion gemcitabine with vs without oxaliplatin vs standard infusion gemcitabine.
* Compare the toxicity of these regimens in these patients.
* Compare the objective response in patients treated with these regimens.
* Compare the patterns of failure and progression-free survival of patients treated with these regimens.
* Compare the reported frequency of deep vein thrombosis and pulmonary embolism among patients treated with these regimens.
* Compare the changes in quality of life, including improved symptom control and/or additional side effects of patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to ECOG performance status (0 or 1 vs 2) and disease stage (locally advanced vs metastatic). Patients are randomized to 1 of 3 treatment arms.

* Arm I (standard treatment): Patients receive gemcitabine IV over 30 minutes once weekly for 7 weeks followed by 1 week of rest for course 1 only. In all subsequent courses, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15, with courses repeating every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 150 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive gemcitabine IV over 100 minutes on day 1 and oxaliplatin IV over 120 minutes on day 2. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then at 8 and 16 weeks.

Patients are followed for 3 years.

PROJECTED ACCRUAL: A total of 789 patients (263 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced or metastatic pancreatic adenocarcinoma or poorly differentiated carcinoma
* Ineligible for curative resection
* Measurable and/or nonmeasurable disease
* Must have evidence of disease outside prior radiation fields OR radiologically confirmed progression of disease within the radiation fields after completion of radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,500/mm^3 OR
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 125,000/mm^3

Hepatic

* Bilirubin < 2.0 mg/dL
* AST < 3 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No uncontrolled cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test

  * Negative vaginal ultrasound for patients with an elevated beta human chorionic gonadotropin level
* Fertile patients must use effective nonhormonal contraception
* No other malignancies within the past 5 years except nonmetastatic, nonmelanoma skin cancer, carcinoma in situ of the cervix, or cancer cured by surgery or small field radiotherapy
* No active or uncontrolled infection
* No other active illness that would preclude study participation
* No symptomatic sensory peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for metastatic disease
* No prior (including adjuvant) gemcitabine or oxaliplatin
* Prior adjuvant chemotherapy allowed provided there was more than 6 months between the last dose of adjuvant chemotherapy and recurrence of pancreatic cancer
* Prior chemotherapy as a radiosensitizing agent allowed* NOTE: *To the primary site

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy to the primary tumor site and recovered
* No prior radiotherapy to more than 25% of the functional bone marrow

Surgery

* See Disease Characteristics
* Prior surgical resection allowed

Other

* No concurrent participation in supportive care trials
* Concurrent enrollment on protocol ECOG-E1Y03 allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Poplin, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (61):
- United States (60):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Medical Center of Aurora - South Campus, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers - Denver Rose, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - La Grange Oncology Associates, La Grange, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Poplin E, Feng Y, Berlin J, Rothenberg ML, Hochster H, Mitchell E, Alberts S, O'Dwyer P, Haller D, Catalano P, Cella D, Benson AB 3rd. Phase III, randomized study of gemcitabine and oxaliplatin versus gemcitabine (fixed-dose rate infusion) compared with gemcitabine (30-minute infusion) in patients with pancreatic carcinoma E6201: a trial of the Eastern Cooperative Oncology Group. J Clin Oncol. 2009 Aug 10;27(23):3778-85. doi: 10.1200/JCO.2008.20.9007. Epub 2009 Jul 6. PMID 19581537
- [Result] Liebes L, Levy DE, Poplin E, et al.: Gemcitabine (G) plasma and intracellular pharmacokinetics in E6201: greater metabolite levels using fixed dosing rate (FDR) delivery. [Abstract] J Clin Oncol 24 (Suppl 18): A-2024, 2006.
- [Result] Poplin E, Levy DE, Berlin J, et al.: Phase III trial of gemcitabine (30-minute infusion) versus gemcitabine (fixed-dose-rate infusion[FDR]) versus gemcitabine + oxaliplatin(GEMOX) in patients with advanced pancreatic cancer (E6201). [Abstract] J Clin Oncol 24 (Suppl 18): A-LBA4004, 180s, 2006.